CLINICAL TRIAL: NCT05466656
Title: SUMAMOS EXCELENCIA Project: Assessment of Implementation of Best Practices in a National Health System (Second Edition)
Brief Title: Sumamos Excelencia 2022
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Teresa Moreno Casbas (Other Government)
Collaborators: The Spanish Centre for Evidence Based Nursing and Healthcare (Unknown)
Responsible Party: Sponsor-Investigator, Teresa Moreno Casbas, Director of the Nursing and helathcare research Unit (Investén-isciii), Instituto de Salud Carlos III
Organization: Instituto de Salud Carlos III (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SE_CECBE_2022
Record Dates: First submitted 2022-07-15; First posted 2022-07-20 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Pain; Incontinence, Urinary; Obesity, Childhood; Breastfeeding
Keywords: Implementation Science; Evidence-Based Practice; Evidence-Based Nursing; Nursing Care; Quality of Health Care; Clinical Audit
MeSH Terms: conditions — Pain; Urinary Incontinence; Pediatric Obesity; Breast Feeding

STUDY DESIGN:
Intervention Model Description: Quasi-experimental, uncontrolled, before-and-after study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Quasi-experimental uncontrolled, before-and-after. (Experimental): The intervention will consist of the use of a continuous quality improvement cycle model and implementation of its strategies in clinical practice, according to the study unit in question and the scope of action.
  Interventions: Other: Continuous quality improvement cycle model

INTERVENTIONS:
Other: Continuous quality improvement cycle model — The continuous quality improvement cycle model consist in a process of improvement by reference to a prior baseline clinical audit. It implies a local situation analysis, identifying barriers to improvements in clinical practice, and drawing up and implementing a plan of action for improving adherence to pre-established criteria. The goal is to establish interprofessional processes within the teams, in order to: examine the barriers that hinder the use of evidence in fostering best practices; and contribute to the development of implementation programmes for overcoming such obstacles.

SUMMARY:
There is a gap between research and clinical practice, leading to variability in decision-making. Clinical audits are an effective strategy for improving implementation of best practices. Quasi-experimental, multicentre, before and after. Primary care, hospital units and nursing homes, and the patients attended at both. Implementation of evidence-based recommendations by application of a continuous quality improvement cycle model (process of improvement by reference to a prior baseline clinical audit. Data will be collected at baseline and, during the first year of follow up, at months (3, 6, 12)

DETAILED DESCRIPTION:
Aim: To assess the effectiveness of implementing evidence-based recommendations using a continuous quality improvement cycle model on patient outcomes and healthcare quality. Design: Quasi-experimental, multicentre, before-and-after. Methods: NHS units and Nursing Homes, patients attended by them and professionals implementing the recommendations. Intervention: implementation of evidence-based recommendation with a continuous quality improvement cycle's model (process of improvement by reference to a prior baseline clinical audit). Variables: Process and outcome criteria with respect to assessment and management of pain, management of urinary incontinence, prevention of child obesity, promotion of breastfeeding, promotion of hand hygiene, competencies in evidence-based practice, barriers to the implementation and strategies for overcoming them. Data will be collected at baseline and, during the first year of follow-up, at months 3, 6 and 12, with data on patients and indicators being drawn from clinical histories and records. Descriptive analysis and comparison of the effectiveness of the intervention by means of inferential analysis and analysis of trends across follow-up. 95% confidence level. This project is partially funded by The Spanish Centre for Evidence Based Nursing and Healthcare. Project duration 2022-2024.

This project is a second edition of The SUMAMOS EXCELENCIA Project: Assessment of Implementation of Best Practices in a National Health System (NCT03725774), with a similar design but with changes in some of the themes.

ELIGIBILITY:
Inclusion Criteria:

1. Unit inclusion criteria:

   * NHS units and nursing homes which voluntary adhere to the project.
   * NHS units and nursing homes providing direct patient care and commit to implement evidence-based recommendations on hand hygiene and one of the following topics: pain assessment and management, urinary incontinence management, obesity prevention and breastfeeding promotion. For the purposes of this study, a "unit" is defined as any service, centre or institution that delivers health services to a homogeneous group of patients who share similar characteristics.
2. Patient inclusion criteria: The study will include all patients attended in the units participating in the study, who meet the following criteria, depending on the recommendations to be implemented in each unit:

   1. Pain:

      * People susceptible to suffering some type of pain regardless of age.
      * Patients treated in acute or chronic health institutions (Hospitals, Nursing Homes or Primary Care).
   2. Urinary incontinence:

      * Patients 18 years or older.
      * Patients with uncomplicated stress, urge or mixed urinary incontinence
      * At least 7 days of admission or possibility of continuity of care preferably up to 6 weeks.
   3. Obesity:

      * Babies and preschool children up to 12 years old.
      * For ages 2 to 12 years (inclusive), children must not be overweight or obese 1 year prior to baseline measurement (in February 2021 or at the closest review to February 2021 at which BMI is recorded).
      * Good general health.
   4. Breastfeeding:

      * Lactating people.
      * Healthy neonates of gestational age greater than 36 weeks, with birth weight greater than or equal to 2500 gr.
      * Couples and relatives within the support network.
      * Postpartum period and up to 6 months of life of the baby (183 days of life, included).
      * In primary care, only non-urgent care will be included.
   5. Hand hygiene:

      * All health professionals who care for patients in the units participating in the study.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Urinary incontinence assessment | 15 months
  Assessment of presence of urinary incontinence. Total number of patients in whom the presence of urinary incontinence has been initially assessed, and who are registered / Total number of patients with positive detection of urinary incontinence during the data collection period) * 100
Voiding diary | 15 months
  Record of all urination and leakage for 3 consecutive days. (Total number of patients with a voiding diary of 3 days recorded / Total number of patients with urinary incontinence discharged or attended during the data collection period) * 100
Scheduled urination | 15 months
  Using verbal and physical prompts or signals to make people pay attention to their dry/wet situation and the need to go to the bathroom. (Total number of patients with a scheduled urination care plan, and it is registered / Total number of patients with urinary incontinence and a 3-day voiding diary discharged or attended in the data collection period) * 100
Bladder training | 15 months
  Program of education and programmed evacuation in which the intervals of micturition are gradually adjusted. (Total number of patients with a bladder training care plan, and it is registered / Total number of patients with urinary incontinence and a 3-day voiding diary discharged or attended in the data collection period) * 100
Pelvic floor exercises | 15 months
  The individualized education and training of pelvic floor exercises. (Total number of patients with a pelvic floor exercise care plan, and it is registered / Total number of patients with urinary incontinence and a 3-day voiding diary discharged or attended in the data collection period) * 100
Severity | 15 months
  Severity of urinary incontinence. Total number of patients with different levels of urinary incontinence 24 hours prior to assessment / Total number of patients with urinary incontinence during the data collection period) x 100
Impact | 15 months
  Impact of urinary incontinence. (Total number of patients whose urinary incontinence has an impact on their quality of life, in the 24 hours prior to the assessment / Total number of patients with urinary incontinence during the data collection period) x 100
Improvement | 15 months
  Perception of improvement in urinary incontinence. (Total number of patients who perceive an improvement 6 weeks after the intervention / Total number of patients with urinary incontinence before the start of the intervention) x100
Detection of pain at admission | 15 months
  Detection of pain at admission. (Total number of patients in whom pain detection was performed upon admission or at the start of care, and it is registered / Total number of patients discharged or attended in the collection period data) x100
Pain related to a procedure likely to cause pain | 15 months
  Detection of pain related to a procedure likely to cause pain. This indicator evaluates whether the assessment of pain linked to the painful procedure is carried out before and after the procedure, it is also recommended to assess pain during the procedure in cases where it is possible. (Total number of patients in whom pain has been detected after a procedure likely to cause pain, and is registered / Total number of patients in whom a procedure likely to cause pain has been performed in the data collection period data) x100
Pain after a change in the patient's clinical situation | 15 months
  Detection of pain after a change in the patient's clinical situation (clinical situation: significant clinical change, in the general condition of the patient or in their pain, which requires the referral of the patient to a professional with the skills to resolve it). (Total number of patients in whom pain has been detected after a change in their clinical situation, and it is registered / Total number of patients with a change in their clinical situation in the data collection period) x100
Pain intensity assessment | 15 months
  Pain assessment measured with a pain intensity assessment tool. (Total number of patients who have an assessment of pain intensity, and it is recorded / Total number of patients with positive detection of pain in the data collection period) x100
Comprehensive pain assessment | 15 months
  Comprehensive pain assessment takes into account various factors related to pain, including: location of pain, circumstances related to the onset of pain, type of pain, pain intensity, associated symptoms, effect of pain on activities, effect of pain on patient rest and sleep, treatment, relevant medical history, factors that influence pain management. To be considered a comprehensive assessment, at least 60% of the 10 criteria must be performed and recorded. (Total number of patients who have done a comprehensive pain assessment, and it is registered / Total number of patients with positive pain detection in the data collection period) x100
Pain management care plan | 15 months
  Establishing and implementing a pain management care plan for the patient based on the results of the person's assessment, which would include: pharmacological and non-pharmacological measures, the person's goals and appropriate and effective pain management strategies. (Total number of patients with a care plan for acute or chronic pain, and it is registered / Total number of patients with positive detection of pain or susceptible to have pain in the data collection period) x100
Patient or/and caregiver education on pain | 15 months
  Patient or/and caregiver education on the importance of communicating pain, pharmacological, physical and psychological pain management options, how to take the analgesic medication, manage the possible side effects and how the follow-up will be done and who can be consulted with possible doubts. (Total number of patients, family members or caregivers who have received education on pain management, at least once during the care process, and it is registered / Total number of patients with positive detection of pain or likely to have pain in the data collection period) x100
Intensity of pain on admission or in the first 24 hours after surgery or at the start of care | 15 months
  Intensity of pain on admission or in the first 24 hours after surgery or at the start of care measured in numerical format, with the value that corresponds to the scale used in the unit for the assessment of pain, units must indicate on the form the scale they have used. (Sum of pain intensity of patients with positive pain detection or likely to have pain / Total number of patients with assessed pain intensity in the data collection period)
Maximum pain | 15 months
  Maximum scored reported by patients and registered by nurses after pain intensity assessment using an assessment tool. Units must indicate on the form the assessment tool they have used. (Sum of the maximum intensity of pain during the stay or care of patients with positive detection of pain or likely to have pain / Total number of patients with pain intensity assessed in the data collection period)
Skin-to-skin contact | 15 months
  Skin-to-skin contact is the placement of a newborn, naked or with a diaper and cap, in a prone position on the bare chest of a person, covered with a previously heated blanket to prevent heat loss. It should be facilitated immediately (up to 1 hour) after birth or once the child and the nursing person are clinically stable. (Number of infants performing skin-to-skin immediately after birth or with clinically stable dyad /Total number of infants) x100 Dyad: A couple formed by the mother and the nursing baby who form a bond with each other.
Postpartum assessment of breastfeeding | 15 months
  Assessment of breastfeeding completed within the first 24 hours of the newborn life. The objective is that in the first 24 hours the breastfeeding person is able to identify: proper position and grip, efficient breast milk transfer, support networks, breastfeeding self-efficacy, risks of mood disorders, assessment of the newborn in relation to breastfeeding. To carry out the assessment, a breastfeeding assessment tool may be used. (Number of dyads assessed on the breastfeeding process in the first 24 hours/Total number of dyads) x100 Dyad: A couple formed by the mother and the nursing baby who form a bond with each other.
Assessment of breastfeeding after the first 24 hours and before discharge | 15 months
  Assessment of breastfeeding completed after first 24 hours of the newborn life and before hospital discharge. The objective is that before hospital discharge the breastfeeding person is able to identify: proper position and grip, efficient breast milk transfer, support networks, breastfeeding self-efficacy, risks of mood disorders, assessment of the newborn in relation to breastfeeding. To carry out the assessment, a breastfeeding assessment tool may be used. (Number of dyads assessed on the breastfeeding process after the first 24 hours and before hospital discharge / Total number of dyads) x100 Dyad: A couple formed by the mother and the nursing baby who form a bond with each other.
Early assessment of breastfeeding in primary care | 15 months
  In Primary Care, early assessment is considered completed between birth and day 8 of the neonate's life (included). To carry out the assessment, a breastfeeding assessment tool may be used. (Number of dyads assessed early on the process of breastfeeding (between birth and 8 days of life / Total number of dyads between birth and 8 days of life of the newborn) x 100 Dyad: A couple formed by the mother and the nursing baby who form a bond with each other.
Follow-up assessment of breastfeeding in primary care (from 9 days of life to 6 months) | 15 months
  In Primary Care, the follow-up evaluation is carried out between 9 days of life and 6 months/183 days of life of the neonate (included). To carry out the assessment, a breastfeeding assessment tool may be used. (Number of dyads assessed on the breastfeeding process from 9 days of life to 6 months / Total number of dyads from 9 days of life to 6 months of the newborn) x100 Dyad: A couple formed by the mother and the nursing baby who form a bond with each other.
Breastfeeding education for the breastfeeding person | 15 months
  In Hospital Care, it is considered completed if postpartum training has been carried out and resources have been provided to the mother by the interprofessional team in breastfeeding before hospital discharge. In Primary Care, it is considered completed if training has been carried out and resources have been provided to the mother after hospital discharge by the interprofessional team in breastfeeding, at least once in the period after discharge to 8 days or in the period from 9 days to 6 months, in the same visit or in successive visits. (Number of lactating persons receiving education in breastfeeding / Total number of dyads) x100 Dyad: A couple formed by the mother and the nursing baby who form a bond with each other.
Breastfeeding education and support for family members | 15 months
  In hospital care, it is considered completed if education and support in breastfeeding has been carried out for family members before hospital discharge. In Primary Care, it is considered accomplished if breastfeeding education and support has been provided to family members, at least once in the period after discharge to 8 days or in the period from 9 days to 6 months, in the same visit or on successive visits. (Number of dyads whose family has received education and support in breastfeeding / Total number of dyads) x100 Dyad: A couple formed by the mother and the nursing baby who form a bond with each other.
Type of breastfeeding of the newborn during the hospital stay | 15 months
  Type of breastfeeding of the newborn during the hospital stay. (Number of infants exclusively breastfed, receiving mixed breastfeeding or not breastfed during hospital stay / Total number of infants discharged) x100 Exclusive breastfeeding: The infant receives directly or indirectly breast milk. He does not receive any other type of solid or liquid food.
  Mixed breastfeeding: The infant receives breast milk as well as other solid and liquid foods (including water), including non-human milk or formula.
  Non-breastfeeding: The infant receives artificial milk and/or animal milk. The infant does not receive breast milk.
Type of breastfeeding of the newborn in early stage | 15 months
  Type of breastfeeding of the newborn from birth to 8 days of life assessed in Primary care. (Number of newborns who were exclusively breastfed, received mixed breastfeeding or were not breastfed from birth to 8 days of life / Total number of newborns between 0 and 8 days of life) x100 Exclusive breastfeeding: The infant receives directly or indirectly breast milk. He does not receive any other type of solid or liquid food.
  Mixed breastfeeding: The infant receives breast milk as well as other solid and liquid foods (including water), including non-human milk or formula.
  Non-breastfeeding: The infant receives artificial milk and/or animal milk. The infant does not receive breast milk.
Type of breastfeeding of the newborn in follow-up 1 | 15 months
  Type of breastfeeding of the newborn from 9 to 90 days of life, assessed in Primary Care. (Number of infants exclusively breastfed, receiving mixed breastfeeding or not breastfed from 9 days to 90 days of life / Total number of infants from 9 to 90 days of life) x100 Exclusive breastfeeding: The infant receives directly or indirectly breast milk. He does not receive any other type of solid or liquid food.
  Mixed breastfeeding: The infant receives breast milk as well as other solid and liquid foods (including water), including non-human milk or formula.
  Non-breastfeeding: The infant receives artificial milk and/or animal milk. The infant does not receive breast milk.
Type of breastfeeding of the newborn in follow-up 2 | 15 months
  Type of breastfeeding of the newborn from 91 to 182 days of life assessed in Primary care (Number of newborns who received exclusive breastfeeding, receiving mixed breastfeeding or not breastfed from 91 days to 182 days of life / Total number of newborns from 91 to 182 days of life) x100 Exclusive breastfeeding: The infant receives directly or indirectly breast milk. He does not receive any other type of solid or liquid food.
  Mixed breastfeeding: The infant receives breast milk as well as other solid and liquid foods (including water), including non-human milk or formula.
  Non-breastfeeding: The infant receives artificial milk and/or animal milk. The infant does not receive breast milk.
Exclusive breastfeeding at 6 months | 15 months
  Number of newborns who received exclusive breastfeeding on day 183 of life (Number of newborns who received exclusive breastfeeding on day 183 of life / Total number of newborns with 183 days completed) x100
Training of health professionals | 15 months
  Number of health professionals who have received advanced training and/or continuing education in breastfeeding. The training must have a minimum of 18 hours and include theoretical training and practical application of skills. (Number of health professionals who have received advanced training and/or continuing education in breastfeeding / Total number of health professionals) x100
Assessment to prevent obesity | 15 months
  At least one comprehensive assessment including the assessment of nutrition, physical activity, sedentary behaviour, growth and family environment has been completed in infants from birth to 12 years of age. (Total number of children from birth to 12 years of age who have undergone a comprehensive assessment to prevent obesity, and are registered / Total number of children from birth to 12 years of age with one or more well-child follow-up visits in the previous year) x100
Education and support for parents/primary caregivers | 15 months
  Parents or primary caregivers have received education and support including: breastfeeding, role modelling, children's eating practices, family physical activity, screen time, physical activity, healthy eating; and it is documented. (Total number of children from birth to 12 years of age whose parents or caregivers have received education to promote healthy eating or physical activity habits, by child's age, and is registered / Total number of children from birth to 12 years with one or more well-child follow-up visits in the previous year) x100
Exclusive breastfeeding, children from birth to 6 months of age | 15 months
  Children from 0 to 183 days inclusive who have received exclusive breastfeeding, directly from the breast or stored. (Number of children 0-6 months (or-183 days) who received EXCLUSIVE breastfeeding in the previous 24 hours, and is registered / Total number of children 0-6 months with one or more visits well-infant-child follow-up in the previous year) x100
Breastfeeding, children from 6 months of age up to 2 years | 15 months
  Children with more than 183 days of life who received breastfeeding directly from the breast or stored. (Number of children >6 months and up to 2 years (more than 183 days-2 years) who received breastfeeding in the previous 24 hours, and is registered / Total number of children >6 months - and up 2 years with one or more well-infant-child follow-up visits in the previous year) x100
Sedentary behaviour | 15 months
  Number of children from birth to 12 years old who spent the recommended time for their age in front of a screen. (Number of children from birth to 12 years old, whose daily screen time is the recommended for their age, as of parents' declaration, and is registered / Total number of children from births up to 12 years of age with one or more follow-up visits to the well-child infant in the previous year, with assessment of screen time or comprehensive assessment) x100
Daily physical activity | 15 months
  Number of children from birth to 12 years of age who meet the recommendations on amount of daily physical activity. (Number of children from birth to 12 years of age who meet the recommendations on amount of daily exercise, and are registered / Total number of children from birth to 12 years of age with one or more follow-up visits of the healthy infant-child in the previous year, with assessment of physical activity or comprehensive assessment) x100
Incidence of childhood obesity | 15 months
  Incidence of childhood obesity. (Number of children between 2 and 12 years old (included) whose BMI for their age exceeds the percentile to be considered obese according to WHO standards, at the LAST follow-up VISIT of the infant/well-child, and is registered / Number of children between 2 and 12 years of age (included) with one or more well-child infant follow-up visits in the previous year, whose BMI has been assessed in the measurement period) x100
ICU beds with alcohol-based preparations at the point of care | 15 months
  Availability of the alcohol-based preparations in the Intensive Care Units (Hospital care) as close as possible to the place where an activity that requires contact with the patient and/or their immediate environment is going to be carried out and without having to leave the patient's area. Point of care is the place where the patient, the health professional and the care or treatment that involves contact with the patient coincide. (Number of ICU beds in the unit, with base alcoholic preparations at the point of care / Number of ICU beds in the unit) x100
Hospital beds with alcohol-based preparations at the point of care | 15 months
  Availability of the alcohol-based preparations in the hospital units (excluding ICU beds) as close as possible to the place where an activity that requires contact with the patient and/or their immediate environment is going to be carried out and without having to leave the patient's area. Point of care is the place where the patient, the health professional and the care or treatment that involves contact with the patient coincide. (Number of hospitalization beds in the unit, with alcohol-based preparations at the point of care)/(Number of beds in the unit) x100
Consumption of alcohol-based preparations in hospitalization | 15 months
  Litres of alcohol-based preparations consumed in hospitalization units with admission, including ICU (Number of litres of alcohol-based preparations delivered / Total number of stays in the evaluated period) x1000 Total number of stays in the evaluated period: It refers to the stays of hospitalized patients, where stay = Date of discharge - Date of admission, during the indicator calculation period.
Consumption of alcohol-based preparations in Primary Care centers | 15 months
  Litres of alcohol-based preparations consumed in primary care centres. (Number of liters of alcohol-based preparations delivered in primary care / Total number of consultations in the evaluated period) x10000
Consumption of alcohol-based preparations in hospital units without admission | 15 months
  Litres of alcohol-based preparations consumed in hospital units without admission (outpatient consultations, day hospital, etc.). (Number of liters of alcohol-based preparations@delivered in a hospital unit without admission / Total number of consultations in the evaluated period) x1000
Consumption of alcohol-based preparations in Nursing Homes. | 15 months
  Litres of alcohol-based preparations consumed in Nursing Homes (Number of liters of alcohol-based preparations delivered in Nursing Homes / Total number of residents in the evaluated period) x100

SECONDARY OUTCOMES:
Type of institution | 15 months
  Hospital unit, primary care unit or nursing home unit.
Size of hospital unit | 15 months
  Average number of admissions received per year.
Size of Nursing home | 15 months
  Total number of beds in the nursing home unit.
Size of primary care unit | 15 months
  Average number of appointments per day in the units.
No. Nurses | 15 months
  Total number of nurses working in the unit by November 2021.
No. Healthcare assistants | 15 months
  Total number of healthcare assistants working in the unit by November 2021.
Type of unit | 15 months
  Age, health problems and care required by the patients attended by the unit on a regular basis.
Date of discharge | 15 months
  Patients discharge date in case of hospital admissions.
Date of attention | 15 months
  Date when patients were attended in case of primary care.
Date of residence | 15 months
  Date when patients were a resident in case of socio-healthcare centres.
Age | 15 months
  Age of patients.
Sex | 15 months
  Sex of patients.
Mother´s age | 15 months
  Age of the mother.
Breastfeeding for the first time | 15 months
  First time the mother is facing breastfeeding or not.
Type of birth | 15 months
  Way in which the newborn was born: vaginal delivery, instrumental birth, caesarean section.
Weeks of gestation | 15 months
  Number of weeks of pregnancy.
Weight at birth | 15 months
  Weight of the newborn at birth, measured in grams.
Child weight | 15 months
  Child's weight measured in kilograms.
Size | 15 months
  Height: child's height measured in centimetres.
Reason for admission/consultation | 15 months
  Reason for admission/consultation of patients. Reason for the patient to be admitted to the Hospital or to attend the consultation.
Past-medical history | 15 months
  History of previous illness, surgery or painful experiences of the patient.
Barriers | 15 months
  Barriers for the implementation of evidence-based recommendations in the units assessed using a questionnaire adapted from the TICD checklist.
EBP competencies | 15 months
  Competencies in evidence-based practice of the healthcare professionals working in the units that are implementing evidence-based recommendations, assessed with the questionnaire EBP-COQ Prof©.

CONTACTS AND LOCATIONS:
Overall Officials: María Teresa Moreno-Casbas, Doctor, Study Director — Instituto de Salud Carlos III; Esther González-María, Doctor, Principal Investigator — Instituto de Salud Carlos III; Leticia Bernués-Caudillo, PhD Candidate, Study Chair — Instituto de Salud Carlos III; Candela Cameselle-Lago, PhD Candidate, Study Chair — Instituto de Salud Carlos III; Laura Albornos-Muñoz, PhD Candidate, Study Chair — Instituto de Salud Carlos III
Locations (1):
- Instituto de Salud Carlos III - Unidad de Investigación en Cuidados y Servicios de Salud, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kreindler SA. What if implementation is not the problem? Exploring the missing links between knowledge and action. Int J Health Plann Manage. 2016 Apr;31(2):208-26. doi: 10.1002/hpm.2277. Epub 2014 Nov 25. PMID 25424863
- [Background] Morris ZS, Wooding S, Grant J. The answer is 17 years, what is the question: understanding time lags in translational research. J R Soc Med. 2011 Dec;104(12):510-20. doi: 10.1258/jrsm.2011.110180. PMID 22179294
- [Background] Squires JE, Estabrooks CA, Gustavsson P, Wallin L. Individual determinants of research utilization by nurses: a systematic review update. Implement Sci. 2011 Jan 5;6:1. doi: 10.1186/1748-5908-6-1. PMID 21208425
- [Background] Meijers JM, Janssen MA, Cummings GG, Wallin L, Estabrooks CA, Y G Halfens R. Assessing the relationships between contextual factors and research utilization in nursing: systematic literature review. J Adv Nurs. 2006 Sep;55(5):622-35. doi: 10.1111/j.1365-2648.2006.03954.x. PMID 16907795
- [Background] Ortuno-Soriano I, Munoz-Jimenez D, Moreno-Casbas T, Albornos-Munoz L, Gonzalez-Maria E; en nombre del Grupo de Trabajo del Programa de implantacion de buenas practicas en Centros Comprometidos con la Excelencia en Cuidados(R). Evaluation of implementation strategies of the Best Practices Spotlight Organisations (BPSO) Project in Spain. Enferm Clin (Engl Ed). 2020 May-Jun;30(3):222-230. doi: 10.1016/j.enfcli.2019.10.027. Epub 2020 May 7. English, Spanish. PMID 32389600
- [Background] Powell BJ, Fernandez ME, Williams NJ, Aarons GA, Beidas RS, Lewis CC, McHugh SM, Weiner BJ. Enhancing the Impact of Implementation Strategies in Healthcare: A Research Agenda. Front Public Health. 2019 Jan 22;7:3. doi: 10.3389/fpubh.2019.00003. eCollection 2019. PMID 30723713
- [Background] Lewis CC, Boyd MR, Walsh-Bailey C, Lyon AR, Beidas R, Mittman B, Aarons GA, Weiner BJ, Chambers DA. A systematic review of empirical studies examining mechanisms of implementation in health. Implement Sci. 2020 Apr 16;15(1):21. doi: 10.1186/s13012-020-00983-3. PMID 32299461
- [Background] Allen P, Pilar M, Walsh-Bailey C, Hooley C, Mazzucca S, Lewis CC, Mettert KD, Dorsey CN, Purtle J, Kepper MM, Baumann AA, Brownson RC. Quantitative measures of health policy implementation determinants and outcomes: a systematic review. Implement Sci. 2020 Jun 19;15(1):47. doi: 10.1186/s13012-020-01007-w. PMID 32560661
- [Background] Moreno-Casbas T. Perspectives: Implementation strategies to adopt and integrate evidence-based nursing. What are we doing? J. Res. Nurs. 2015;20:729-33.
- [Background] Lau R, Stevenson F, Ong BN, Dziedzic K, Treweek S, Eldridge S, Everitt H, Kennedy A, Qureshi N, Rogers A, Peacock R, Murray E. Achieving change in primary care--causes of the evidence to practice gap: systematic reviews of reviews. Implement Sci. 2016 Mar 22;11:40. doi: 10.1186/s13012-016-0396-4. PMID 27001107
- [Background] Almazrou SH, Alfaifi SI, Alfaifi SH, Hakami LE, Al-Aqeel SA. Barriers to and Facilitators of Adherence to Clinical Practice Guidelines in the Middle East and North Africa Region: A Systematic Review. Healthcare (Basel). 2020 Dec 15;8(4):564. doi: 10.3390/healthcare8040564. PMID 33333843
- [Background] Davies B, Edwards N, Ploeg J, Virani T. Insights about the process and impact of implementing nursing guidelines on delivery of care in hospitals and community settings. BMC Health Serv Res. 2008 Feb 2;8:29. doi: 10.1186/1472-6963-8-29. PMID 18241349
- [Background] Ploeg J, Davies B, Edwards N, Gifford W, Miller PE. Factors influencing best-practice guideline implementation: lessons learned from administrators, nursing staff, and project leaders. Worldviews Evid Based Nurs. 2007;4(4):210-9. doi: 10.1111/j.1741-6787.2007.00106.x. PMID 18076464
- [Background] Mickan S, Burls A, Glasziou P. Patterns of 'leakage' in the utilisation of clinical guidelines: a systematic review. Postgrad Med J. 2011 Oct;87(1032):670-9. doi: 10.1136/pgmj.2010.116012. Epub 2011 Jun 29. PMID 21715571
- [Background] Fleiszer AR, Semenic SE, Ritchie JA, Richer MC, Denis JL. A unit-level perspective on the long-term sustainability of a nursing best practice guidelines program: An embedded multiple case study. Int J Nurs Stud. 2016 Jan;53:204-18. doi: 10.1016/j.ijnurstu.2015.09.004. Epub 2015 Sep 8. PMID 26453418
- [Background] Baker R, Camosso-Stefinovic J, Gillies C, Shaw EJ, Cheater F, Flottorp S, Robertson N. Tailored interventions to overcome identified barriers to change: effects on professional practice and health care outcomes. Cochrane Database Syst Rev. 2010 Mar 17;(3):CD005470. doi: 10.1002/14651858.CD005470.pub2. PMID 20238340
- [Background] Flodgren G, Deane K, Dickinson HO, Kirk S, Alberti H, Beyer FR, Brown JG, Penney TL, Summerbell CD, Eccles MP. Interventions to change the behaviour of health professionals and the organisation of care to promote weight reduction in overweight and obese people. Cochrane Database Syst Rev. 2010 Mar 17;(3):CD000984. doi: 10.1002/14651858.CD000984.pub2. PMID 20238311
- [Background] Esposito P, Dal Canton A. Clinical audit, a valuable tool to improve quality of care: General methodology and applications in nephrology. World J Nephrol. 2014 Nov 6;3(4):249-55. doi: 10.5527/wjn.v3.i4.249. PMID 25374819
- [Background] Wentland BA, Hinderer KA. A Nursing Research and Evidence-Based Practice Fellowship Program in a Magnet(R)-designated pediatric medical center. Appl Nurs Res. 2020 Oct;55:151287. doi: 10.1016/j.apnr.2020.151287. Epub 2020 May 15. PMID 32482374
- [Background] Holmes BJ, Best A, Davies H, Hunter D, Kelly MP, Marshall M, Rycroft-Malone J. Mobilising knowledge in complex health systems: A call to action. Evid. Policy 2017;13:539-60.
- [Background] Powell BJ, McMillen JC, Proctor EK, Carpenter CR, Griffey RT, Bunger AC, Glass JE, York JL. A compilation of strategies for implementing clinical innovations in health and mental health. Med Care Res Rev. 2012 Apr;69(2):123-57. doi: 10.1177/1077558711430690. Epub 2011 Dec 26. PMID 22203646
- [Background] Ivers N, Jamtvedt G, Flottorp S, Young JM, Odgaard-Jensen J, French SD, O'Brien MA, Johansen M, Grimshaw J, Oxman AD. Audit and feedback: effects on professional practice and healthcare outcomes. Cochrane Database Syst Rev. 2012 Jun 13;2012(6):CD000259. doi: 10.1002/14651858.CD000259.pub3. PMID 22696318
- [Background] Sinuff T, Muscedere J, Rozmovits L, Dale CM, Scales DC. A qualitative study of the variable effects of audit and feedback in the ICU. BMJ Qual Saf. 2015 Jun;24(6):393-9. doi: 10.1136/bmjqs-2015-003978. Epub 2015 Apr 27. PMID 25918432
- [Background] Munoz Jimenez D. From evidence-based nursing to healthcare practice: The evaluation of results as an integrating element. Enferm Clin (Engl Ed). 2018 May-Jun;28(3):149-153. doi: 10.1016/j.enfcli.2018.04.004. No abstract available. English, Spanish. PMID 29778244
- [Background] Christina V, Baldwin K, Biron A, Emed J, Lepage K. Factors influencing the effectiveness of audit and feedback: nurses' perceptions. J Nurs Manag. 2016 Nov;24(8):1080-1087. doi: 10.1111/jonm.12409. Epub 2016 Jun 16. PMID 27306646
- [Background] GBD 2015 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 310 diseases and injuries, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1545-1602. doi: 10.1016/S0140-6736(16)31678-6. PMID 27733282
- [Background] Duenas M, Salazar A, Ojeda B, Fernandez-Palacin F, Mico JA, Torres LM, Failde I. A nationwide study of chronic pain prevalence in the general spanish population: identifying clinical subgroups through cluster analysis. Pain Med. 2015 Apr;16(4):811-22. doi: 10.1111/pme.12640. Epub 2014 Dec 19. PMID 25530229
- [Background] García FJ, Salinas J, Madurga B, Cózar JM, Esteban M. Guía de atención a personas con incontinencia urinaria [internet]. Madrid: Asociación Española de Urología; Enero 2020 [consultado abril de 2021]. Available in: https://www.consejogeneralenfermeria.org/documentos-de-interes/guias-clinicas/send/67-guias-clinicas/908-guia-de-atencion-a-personas-con-incontinencia-urinaria
- [Background] Dufour S, Wu M. No. 397 - Conservative Care of Urinary Incontinence in Women. J Obstet Gynaecol Can. 2020 Apr;42(4):510-522. doi: 10.1016/j.jogc.2019.04.009. PMID 32303295
- [Background] Estudio ALADINO 2019: Estudio sobre Alimentación, Actividad Física, Desarrollo Infantil y Obesidad en España 2019. Agencia Española de Seguridad Alimentaria y Nutrición. Ministerio de Consumo. Madrid, 2020
- [Background] Departamento de Salud del Gobierno Vasco. Estrategia de prevención de la obesidad infantil en Euskadi. PLAN SANO. 2019. Editado por Servicio Central de publicaciones del Gobierno Vasco. Disponible en: https://www.euskadi.eus/estrategia/prevencion-de-la-obesidad-infantil-en-euskadi/web01-a2osabiz/es/
- [Background] World Health Organization. Infant and young child feeding. Ginebra: WHO; 2021 [acceso12/11/2021]. Disponible en: https://www.who.int/news-room/fact-sheets/detail/infant-and-young-child-feeding.
- [Background] Encuesta Nacional de Salud de España 2017. Instituto nacional de estadística. [acceso 25/08/2019]. Disponible en https://www.mscbs.gob.es/estadEstudios/estadisticas/encuestaNacional/encuesta2017.htm
- [Background] OMS, Ministerio de Sanidad. La higiene de las manos en la asistencia ambulatoria y domiciliaria y en los cuidados de larga duración. Guía de aplicación de la estrategia multimodal de la OMS para la mejora de la higiene de las manos y del modelo "Los cinco momentos para la higiene de las manos". Ginebra: Organización Mundial de la Salud. 2013
- [Background] Agencia Española del Medicamento y Producto Sanitarios. Programa Higiene de manos del SNS. Informe de indicadores 2019. Madrid. 2020
- [Background] Estudio nacional de vigilancia de infección nosocomial en servicios de medicina intensiva. Vall d'hebron. Barcelona; 2019. Disponible en: https://hws.vhebron.net/envin-helics/
- [Background] Estudio APEAS. Estudio sobre la seguridad de los pacientes en atención primaria de salud. Madrid: Ministerio de Sanidad y Consumo; 2008.
- [Background] Flottorp SA, Oxman AD, Krause J, Musila NR, Wensing M, Godycki-Cwirko M, Baker R, Eccles MP. A checklist for identifying determinants of practice: a systematic review and synthesis of frameworks and taxonomies of factors that prevent or enable improvements in healthcare professional practice. Implement Sci. 2013 Mar 23;8:35. doi: 10.1186/1748-5908-8-35. PMID 23522377
- [Background] Escobar-Aguilar G, Moreno-Casbas MT, Gonzalez-Maria E, Martinez-Gimeno ML, Sanchez-Pablo C, Orts-Cortes I. The SUMAMOS EXCELENCIA Project. J Adv Nurs. 2019 Jul;75(7):1575-1584. doi: 10.1111/jan.13988. Epub 2019 Apr 2. PMID 30816569
- [Background] Martinez-Gimeno ML, Fernandez-Martinez N, Escobar-Aguilar G, Moreno-Casbas MT, Brito-Brito PR, Caperos JM. SUMAMOS EXCELENCIA(R) Project: Results of the Implementation of Best Practice in a Spanish National Health System (NHS). Healthcare (Basel). 2021 Mar 28;9(4):374. doi: 10.3390/healthcare9040374. PMID 33800670
- See also: website fron the The Spanish Centre for Evidence Based Nursing and Healthcare with the project information — https://evidenciaencuidados.es/